CLINICAL TRIAL: NCT06018454
Title: Preimplantation Genetic Testing for Aneuploidy (PGT-A) Counseling for Patients Undergoing in Vitro Fertilization (IVF)
Brief Title: Preimplantation Genetic Testing for Aneuploidy Counseling
Acronym: PGT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyup Hakan Duran (Other)
Responsible Party: Sponsor-Investigator, Eyup Hakan Duran, Principal investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202208644
Record Dates: First submitted 2023-08-01; First posted 2023-08-30 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Patient Education
MeSH Terms: interventions — Genetic Counseling

STUDY DESIGN:
Intervention Model Description: Patients randomized with computer generated block randomization of ratio 1:1:1 to randomize women to either 10 minute genetic counseling intervention with handout, handout, or no interventions. Randomization allocation will be performed prior to study initiation through the Institute for Clinical and Translational Science (ICTS) via REDCap software.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Provider counseling with pre-test (No Intervention): Counseling regarding PGT-A only with a provider(current standard of care), pre-test provided.
- Handout on PGT-A and provider counseling with pre-test (Experimental): Counseling regarding PGT-A with a provider and review of a handout(educational intervention), pre-test provided.
  Interventions: Other: Handout on PGT-A
- Handout on PGT-A, provider counseling and brief genetic counselor counseling with pre-test (Experimental): Counseling regarding PGT-A only with a provider, review of a handout(educational intervention) and genetic counseling (counseling intervention), pre-test provided.
  Interventions: Other: Handout on PGT-A; Other: Handout on PGT-A and genetic counseling

INTERVENTIONS:
Other: Handout on PGT-A — Educational handout on PGT-A
  Arms: Handout on PGT-A and provider counseling with pre-test; Handout on PGT-A, provider counseling and brief genetic counselor counseling with pre-test
Other: Handout on PGT-A and genetic counseling — Handout on PGT-A and genetic counseling session with a genetic counselor on PGT-A
  Arms: Handout on PGT-A, provider counseling and brief genetic counselor counseling with pre-test

SUMMARY:
Purpose: To evaluate preimplantation genetic testing counseling interventions on patients undergoing in vitro fertilization treatment.

Preimplantation genetic testing for aneuploidy (PGT) allows patients undergoing in vitro fertilization (IVF) to screen embryos for genetic disorders. Preimplantation genetic testing for aneuploidy (PGT-A) is the testing most commonly ordered, and it screens for whole chromosome and large partial chromosome duplications or deletions. Currently, patient counseling varies based on the clinic, ranging from appointments to group seminars with a genetic counselor (GC), geneticist or reproductive endocrinology and infertility (REI) physicians for education regarding PGT. Patient knowledge regarding PGT has been varied with some studies indicating sufficient knowledge, while other studies have shown a potential lack of knowledge. One study indicated a third of patients had regret regarding their decision of whether or not to use PGT-A during IVF and another study indicated patients who choose to undergo PGT did so for reasons that were not evidence based. Additionally, educational materials have been illustrated to be inconsistent and with inappropriate literacy in regards to PGT counseling. One study has shown the potential of improvement with written intervention amongst providers and patients in regards to PGT related to a single genetic condition. The investigators hope to assess the efficacy of PGT-A educational and counseling interventions on patients undergoing IVF.

DETAILED DESCRIPTION:
Procedures: Patients undergoing IVF for the first time will be randomized to one of three groups

1. Provider counseling (current standard care) with pre-test
2. Handout on PGT-A and provider counseling (current standard care + educational intervention) with pre-test
3. Handout on PGT-A, provider counseling and brief genetic counselor counseling (current standard of care + educational and counseling interventions) with pre-test

All patients will receive provider counseling(current standard of care) on PGT-A during their new IVF clinic visit. All groups will take a pre-test on PGT-A prior to receiving provider counseling and (if in an intervention group) prior to receiving handout or handout with brief counseling on PGT-A from a genetic counselor. At the end of their clinic visit, all participants will complete a post-test on PGT-A.

Two weeks after their clinic visit, all participants will receive a 2nd post-test on PGT-A and the SURE questionnaire to assess retained knowledge about PGT-A and decisional conflict about their choice to use PGT-A in their treatment cycle.

As there is not a validated knowledge survey for PGT-A, investigators have developed their own for pre- and post-tests. In order to validate the survey prior to using it in this study, investigators plan to enroll the first 100 participants in a pilot study to validate the instrument. The number needed for validation will depend on how much pilot participants scores vary between pre and post test. Participants in the pilot portion of the study will be asked to complete a pre-test on PGT-A, read the informational handout about PGT-A, and then complete a post test on PGT-A prior to their IVF appointment. Statisticians will analyze the pilot data as received, and will inform investigators when a sufficient number has been reached for survey validation. Once validated, the pilot arm of the study will be closed and will begin enrolling participants in the randomized trial portion described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing in vitro fertilization (IVF)

Exclusion Criteria:

* Patients who have previously undergone IVF would be excluded.
* Patients who have previously discussed PGT with a genetic counselor would be excluded.
* Patients who do not speak English will be excluded.
* Patients who are employees of the clinic would be excluded.
* Patients who have an indication for PGT-M or PGT-SR would be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
PGT-A Knowledge scores | Prior to new IVF visit
  Study team designed 7 item knowledge questionnaire. Lowest score being 0 and highest score being 7.
PGT-A Knowledge scores | Immediately following new IVF visit
  Study team designed 7 item knowledge questionnaire. Lowest score being 0 and highest score being 7.
PGT-A Knowledge scores | Two weeks post IVF visit.
  Study team designed 7 item knowledge questionnaire. Lowest score being 0 and highest score being 7.

SECONDARY OUTCOMES:
Decisional conflict as measured by the SURE questionnaire. | Two weeks post IVF visit.
  A validated questionnaire assessing patient decisional conflict on a scale of 0 to 4. Zero indicating no decisional conflict and 1 or greater indicating increasing levels of decisional conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Prapti Singh, DO, Study Director — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gebhart MB, Hines RS, Penman A, Holland AC. How do patient perceived determinants influence the decision-making process to accept or decline preimplantation genetic screening? Fertil Steril. 2016 Jan;105(1):188-93. doi: 10.1016/j.fertnstert.2015.09.022. Epub 2015 Oct 24. PMID 26474735
- [Background] Lee I, Alur-Gupta S, Gallop R, Dokras A. Utilization of preimplantation genetic testing for monogenic disorders. Fertil Steril. 2020 Oct;114(4):854-860. doi: 10.1016/j.fertnstert.2020.05.045. PMID 33040985
- [Background] Kaing A, Rosen MP, Quinn MM. Perceptions, motivations and decision regret surrounding preimplantation genetic testing for aneuploidy. Hum Reprod. 2020 Sep 1;35(9):2047-2057. doi: 10.1093/humrep/deaa154. PMID 32756971
- [Background] Quinn MM, Juarez-Hernandez F, Dunn M, Okamura RJ, Cedars MI, Rosen MP. Decision-making surrounding the use of preimplantation genetic testing for aneuploidy reveals misunderstanding regarding its benefit. J Assist Reprod Genet. 2018 Dec;35(12):2155-2159. doi: 10.1007/s10815-018-1337-8. Epub 2018 Oct 18. PMID 30334131
- [Background] McGowan ML, Burant CJ, Moran R, Farrell R. Patient education and informed consent for preimplantation genetic diagnosis: health literacy for genetics and assisted reproductive technology. Genet Med. 2009 Sep;11(9):640-5. doi: 10.1097/GIM.0b013e3181ac6b52. PMID 19652605
- [Background] Early ML, Kumar P, Marcell AV, Lawson C, Christianson M, Pecker LH. Literacy assessment of preimplantation genetic patient education materials exceed national reading levels. J Assist Reprod Genet. 2020 Aug;37(8):1913-1922. doi: 10.1007/s10815-020-01837-z. Epub 2020 May 29. PMID 32472448
- [Background] Early ML, Strodel RJ, Lake IV, Ruddy JA, Saba JA, Singh SM, Lanzkron S, Mack JW, Meier ER, Christianson MS, Pecker LH. Acceptable, hopeful, and useful: development and mixed-method evaluation of an educational tool about reproductive options for people with sickle cell disease or trait. J Assist Reprod Genet. 2022 Jan;39(1):183-193. doi: 10.1007/s10815-021-02358-z. Epub 2021 Nov 22. PMID 34806131
- [Derived] Singh P, Summers KM, Chanouha N, Thoeny R, Zorn A, Van Voorhis BJ, Sparks AE, Eapen A, Faro EZ, Pawlak SA, Duran EH. A randomized controlled trial of counseling and educational methods on preimplantation genetic testing for aneuploidy for patients pursuing in vitro fertilization. Fertil Steril. 2025 Nov 15;124(5 Pt 2):964-973. doi: 10.1016/j.fertnstert.2025.06.010. Epub 2025 Jun 14. PMID 40523553